CLINICAL TRIAL: NCT01641302
Title: The Effect of Pneumoperitoneum and Trendelenburg Position on Intracranial Pressure: Ultrasonographic Measurement of Optic Nerve Sheath Diameter
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2012-0287.
Record Dates: First submitted 2012-06-28; First posted 2012-07-16 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Robot-assisted Laparoscopic Prostatectomy Under General Anesthesia

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients undergoing robot-assisted laparoscopic prostatectomy: Patients undergoing robot-assisted laparoscopic prostatectomy under general anesthesia

SUMMARY:
The steep Trendelenburg position and pneumoperitoneum during laparoscopic surgery have the potential to cause an increase of intracranial pressure (ICP). Previous studies have proposed that ultrasonographic measurements of the optic nerve sheath diameter (ONSD) correlate with signs of increased ICP. Therefore, this study is aim to confirm the increased ICP by ultrasonographic measurement of ONSD during laparoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (20-90 years of age) scheduled for undergoing robot-assisted laparoscopic prostatectomy undergoing general anesthesia

Exclusion Criteria:

* Patients with previous history of neurologic disease, carotid disease, transient ischemic attack, ocular disease and ocular surgery

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing robot-assisted laparoscopic prostatectomy under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2012-06; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
ultrasonographic measurement of optic nerve sheath diameter | before anesthesia induction, 10 minutes after anesthesia induction, 30 minutes after steep trendelenburg position and pneumoperitoneum, and 10 minutes after supine position, CO2 desufflation.
  A thick layer of gel is applied on the upper closed eyelid. The linear 13- to 6-MHz ultrasound probe is then placed in the gel, without exerting pressure on the eye. Two measurements are taken for each optic nerve: one in the transverse plane, with the probe being horizontal, and one in the sagittal plane, with the probe being vertical. The final ONSD is the mean of these measurements.

CONTACTS AND LOCATIONS:
Locations (1):
- Associate Professor Department of Anesthesiology and Pain Medicine,, Seoul, Seoul, South Korea